CLINICAL TRIAL: NCT01815268
Title: High Dose Influenza Vaccination and Morbidity & Mortality in U.S. Nursing Homes
Brief Title: High-Dose Influenza Vaccine in Nursing Homes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Insight Therapeutics, LLC (Other)
Collaborators: Brown University (Other); Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GRC75-EXT
Record Dates: First submitted 2013-03-11; First posted 2013-03-21 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Influenza
Keywords: Randomized Controlled Trial; Influenza; Influenza vaccine; Flu Vaccine; Fluzone; HD Fluzone; Nursing Home; Hospitalization; Mortality; Health Care worker vaccination; ADL decline; Effectiveness; Elderly; Morbidity; Nursing Home resident; Frail; Institutionalized; Epidemiology; CDC; US; city
MeSH Terms: conditions — Influenza, Human | interventions — Fluzone High-Dose; Influenza Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- HD Vaccine (Residents) + Free Vaccine (Staff) (Experimental): NH facilities randomized to receive high-dose trivalent influenza vaccine (Fluzone High-Dose) for the residents and provided free SD vaccine (Fluzone) for the staff.
  Interventions: Biological: HD Vaccine; Biological: Free Vaccine
- HD Vaccine (Residents) + Usual Care (Staff) (Experimental): NH facilities randomized to receive high-dose trivalent influenza vaccine (Fluzone High-Dose) for the residents and not provided free vaccine for the staff.
  Interventions: Biological: HD Vaccine; Biological: Usual Care
- SD Vaccine (Residents) + Free Vaccine (Staff) (Active Comparator): NH facilities randomized to receive standard dose influenza vaccine (Fluzone) for the residents and provided free standard dose vaccine (Fluzone) for the staff.
  Interventions: Biological: SD Vaccine; Biological: Free Vaccine
- SD Vaccine (Residents) + Usual Care (Staff) (Active Comparator): NH facilities randomized to receive standard dose influenza vaccine (Fluzone) for the residents and not provided free vaccine for the staff.
  Interventions: Biological: SD Vaccine; Biological: Usual Care

INTERVENTIONS:
Biological: HD Vaccine — Nursing home residents over 65 years are allocated to receive high-dose vaccine. Residents under 65 years are provided standard-dose vaccine.
  Other Names: Fluzone High-Dose
  Arms: HD Vaccine (Residents) + Free Vaccine (Staff); HD Vaccine (Residents) + Usual Care (Staff)
Biological: SD Vaccine — Nursing home residents are allocated to receive standard-dose vaccine.
  Other Names: Fluzone
  Arms: SD Vaccine (Residents) + Free Vaccine (Staff); SD Vaccine (Residents) + Usual Care (Staff)
Biological: Free Vaccine — Nursing home facilities are provided free standard-dose vaccine for their staff.
  Other Names: Fluzone
  Arms: HD Vaccine (Residents) + Free Vaccine (Staff); SD Vaccine (Residents) + Free Vaccine (Staff)
Biological: Usual Care — Nursing home staff will have access to influenza vaccine, per standard of care. No free vaccine provided as part of study.
  Arms: HD Vaccine (Residents) + Usual Care (Staff); SD Vaccine (Residents) + Usual Care (Staff)

SUMMARY:
The purpose of this study is to prospectively evaluate relative effectiveness of high dose influenza vaccine in preventing influenza mortality, hospitalization, and functional decline in a nursing home population in the U.S., compared to the standard dose trivalent seasonal influenza vaccine.

DETAILED DESCRIPTION:
SUMMARY: This nationally representative study samples from estimated 6782 Medicare-certified nursing homes co-located within 50 miles of the 122 cities reporting to Center for Disease Control and Prevention (CDC) weekly influenza surveillance. In total, 1000 facilities will be enrolled for random assignment to either: 1) the licensed high dose (HD) trivalent influenza vaccine (High-Dose Fluzone [HD vaccine]), or 2) the standard dose (SD) trivalent influenza vaccine (Fluzone [SD vaccine]) for their residents. Additionally, half the facilities will receive free SD vaccine for their staff and the remaining facilities will practice usual care (no free vaccine) for staff.

BACKGROUND: Influenza and pneumonia (P&I) are leading infectious causes of hospitalization and mortality in community-dwelling older adults and residents of long-term custodial care facilities or nursing homes (NH), and produce substantial annual health care costs. The elderly incur over 90% of this disease burden and NH residents are especially vulnerable given immune senescence, multimorbidity, and close living quarters. While hospitalization rates for NH residents vary considerably between facilities, most occur during the sixteen weeks of peak influenza activity annually. Influenza vaccination, a mainstay in prevention, is recommended in the U.S. for all individuals six months of age and older. Vaccination associates with reduced rates of stroke, heart attack, hospitalization, and death in non-institutional older adult populations. However, the benefit of influenza vaccine for the elderly in general has been questioned, a salient concern for frail elderly, such as NH residents. Influenza vaccination rates vary substantially between nursing homes. Influenza vaccine response declines with advancing age, indicating the need for a better vaccine.

OBJECTIVES: The primary objective is to estimate the differences in all-cause hospitalization rates during influenza season experienced by long-stay nursing home residents, between facilities using HD vaccine vs. SD vaccine. The secondary objective is to estimate the differences in the likelihood of Activities of Daily Living (ADL) functional decline and mortality rates in the study nursing homes.

ELIGIBILITY:
Inclusion Criteria:

* Long-term care facilities within 50 miles of one of the 122 cities that serve as CDC surveillance sites

Exclusion Criteria:

* Facilities already systematically administering HD vaccine to their residents
* Facilities having fewer than 50 long-stay residents
* Hospital-based facilities
* Facilities with more than 20% of the population under age 65
* Facilities not submitting Minimum Data Set (MDS) data

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 823 (Actual)
Dates: Start 2013-02; Primary Completion 2017-05-15 (Actual); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Hospitalization rate | up to 1 year

SECONDARY OUTCOMES:
Change in activities of daily living (ADL) scores | up to 1 year
Facility-level mortality rate | up to 1 year
Hospitalization rate based on vaccine type and influenza strain | Up to 3 years
Cost difference between vaccine types | up to 3 years
Effect of facility policies on staff vaccination rates | up to 3 years

OTHER OUTCOMES:
Difference in hospitalization claims based on staff vaccination status | up to 1 year
  Effect on clinical outcomes of nursing home residents based on staff vaccine uptake.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Gravenstein, MD, MPH, Principal Investigator — Case Western Reserve University; Vincent Mor, PhD, Principal Investigator — Brown University; Ed Davidson, PharmD, MPH, Principal Investigator — Insight Therapeutics, LLC
Locations (3):
- United States (3):
  - Case Western Reserve University, Cleveland, Ohio
  - Brown University, Providence, Rhode Island
  - Insight Therapeutics, LLC, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gozalo PL, Pop-Vicas A, Feng Z, Gravenstein S, Mor V. Effect of influenza on functional decline. J Am Geriatr Soc. 2012 Jul;60(7):1260-7. doi: 10.1111/j.1532-5415.2012.04048.x. Epub 2012 Jun 21. PMID 22724499
- [Background] Fiore AE, Shay DK, Haber P, Iskander JK, Uyeki TM, Mootrey G, Bresee JS, Cox NJ; Advisory Committee on Immunization Practices (ACIP), Centers for Disease Control and Prevention (CDC). Prevention and control of influenza. Recommendations of the Advisory Committee on Immunization Practices (ACIP), 2007. MMWR Recomm Rep. 2007 Jul 13;56(RR-6):1-54. PMID 17625497
- [Background] DiazGranados CA, Dunning AJ, Kimmel M, Kirby D, Treanor J, Collins A, Pollak R, Christoff J, Earl J, Landolfi V, Martin E, Gurunathan S, Nathan R, Greenberg DP, Tornieporth NG, Decker MD, Talbot HK. Efficacy of high-dose versus standard-dose influenza vaccine in older adults. N Engl J Med. 2014 Aug 14;371(7):635-45. doi: 10.1056/NEJMoa1315727. PMID 25119609
- [Background] Keitel WA, Atmar RL, Cate TR, Petersen NJ, Greenberg SB, Ruben F, Couch RB. Safety of high doses of influenza vaccine and effect on antibody responses in elderly persons. Arch Intern Med. 2006 May 22;166(10):1121-7. doi: 10.1001/archinte.166.10.1121. PMID 16717175
- [Background] Falsey AR, Treanor JJ, Tornieporth N, Capellan J, Gorse GJ. Randomized, double-blind controlled phase 3 trial comparing the immunogenicity of high-dose and standard-dose influenza vaccine in adults 65 years of age and older. J Infect Dis. 2009 Jul 15;200(2):172-80. doi: 10.1086/599790. PMID 19508159
- [Derived] Gravenstein S, Davidson HE, Taljaard M, Ogarek J, Gozalo P, Han L, Mor V. Comparative effectiveness of high-dose versus standard-dose influenza vaccination on numbers of US nursing home residents admitted to hospital: a cluster-randomised trial. Lancet Respir Med. 2017 Sep;5(9):738-746. doi: 10.1016/S2213-2600(17)30235-7. Epub 2017 Jul 20. PMID 28736045
- [Derived] Gravenstein S, Dahal R, Gozalo PL, Davidson HE, Han LF, Taljaard M, Mor V. A cluster randomized controlled trial comparing relative effectiveness of two licensed influenza vaccines in US nursing homes: Design and rationale. Clin Trials. 2016 Jun;13(3):264-74. doi: 10.1177/1740774515625976. Epub 2016 Feb 11. PMID 26908539